CLINICAL TRIAL: NCT02568436
Title: Evaluation of Low-Level Laser Therapy (LLLT) Effectiveness in Accelerating Orthodontic Tooth Movement For Dental Crowding Cases: A Randomized Controlled Clinial Trial
Brief Title: Effect of Low Level Laser Therapy in Accelerating Tooth Movement For Dental Crowding Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-02-2015
Record Dates: First submitted 2015-09-26; First posted 2015-10-05 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Maxillary Crowded Teeth
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Decrowding (No Intervention): Crowded upper incisors will be treated in the conventional manner with a fake irradiation without using low level laser therapy.
- Low Level Laser Therapy (Experimental): Each maxillary incisor will be subjected to low level laser therapy at specific times in order to accelerate tooth movement
  Interventions: Radiation: low level laser therapy

INTERVENTIONS:
Radiation: low level laser therapy — low level laser therapy is intended to accelerate tooth movement
  Arms: Low Level Laser Therapy

SUMMARY:
26 participants from the Orthodontic Department at University of Damascus Dental School will be randomly assigned into two groups. In the experimental group, a low level laser with a wave length of 830 nm, output of 150 mw, energy of 2 j per point and application time of 15 seconds per point will be applied on each tooth of the six upper incisors according to this protocol: the root will be divided into 2 halves; gingival and cervical. Laser will be applied in the center of each half from both the buccal and palatal sides which means 4 application points and a total energy of 8 j per each tooth. Control group will undergo typical orthodontic treatment with the laser device applied the same manner but without being turned on (to get the placebo effect for pain reduction effect). This procedure will be repeated after 3, 7, 14 days and each 15 days from the beginning of the second month till the end of the leveling and alignment stage.

DETAILED DESCRIPTION:
The long time needed for orthodontic treatment is considered one of the biggest obstacles which make patients refuse to undergo treatment. It also has many disadvantages including higher caries rates, gingivitis, and root resorption. It also combined commonly with pain, which reducing patient acceptance and cooperation with treatment.

Low level laser therapy in orthodontic has shown pain-reducing effects with an effect in biomodulation which lead to increased orthodontic tooth movement rate and reducing risk of root resorption.

A recent systematic review states that low level laser therapy has shown efficiency in accelerating orthodontic tooth movement, but there is a need for more studies to determine the best protocols regarding energy and frequency. A review of the literature shows that there is no randomized controlled trails evaluating its efficiency in accelerating orthodontic tooth movement in regard of dental crowding cases, which is the main purpose of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between (16 - 24) years.
2. Moderate crowding (3 - 5) mm in the anterior region of the maxillary dental arch with an irregularity index of (7 mm or more) mm according to Little Index with an indication to extract upper two premolars.
3. All upper teeth are existed (except for third molars).
4. Patients have not undergone previous orthodontic treatment.
5. Patients have not undergone any medical treatment that interfere with orthodontic tooth movement (Cortisone, NSAIDs, …).
6. Patient with good oral hygiene (Plaque Index less than 1).

Exclusion Criteria:

1. Any medical condition affecting orthodontic tooth movement.
2. Bad oral hygiene (Plaque Index greater than 1).
3. Any peri-apical lesions developed during treatment.
4. Patient lack of commitment toward follow-up appointments.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Overall Leveling and Alignment Time (OLAT) | This will be measured once the leveling and alignment stage of the orthodontic treatment is finished. This will be measured in days from the commencement of treatment till the final day of leveling and alignment.
  As mentioned above
Change in Leveling and Alignment Improvement Percentage (LAIP) | this outcome will be measured after one month (T1) and two months (T2) of treatment commencement (T0), and at the end of leveling and alignment stage (T3) using Little irregularity index (LII)
  LAIP will be measured by dividing the amount of change in LII value at a specific time intervals (i.e. T3-T0, T2-T0, T1-T0; calculated by subtracting LII value at T1, T2 and T3 from LII value at (T0) by LII value at T0 (i.e. the beginning of treatment).

SECONDARY OUTCOMES:
Change of levels of pain | Using a visual analog scale (VAS), pain will be measured after 1, 6, 24, 48, 72 hours of applying the laser therapy and at 7 days of follow-up.
  Using a visual analog scale, each patient will indicate the severity of his/her perceived pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Moaffak Al-Sayed Hasan, DDS, Principal Investigator — MSc student at the Orthodontic Department, University of Damascus Dental School; Kinda Sultan, DDS MSc PhD, Study Director — Senior Lecturer in Orthodontics, University of Damascus Dental School, SYRIA; Omar Hamadah, DDS MSc PhD, Study Director — Senior Lecturer, Oral Medicine Department, University of Damascus Dental School, Damascus, Syria
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Rif-dimashq Governorate, Syria

REFERENCES:
- [Background] Cruz DR, Kohara EK, Ribeiro MS, Wetter NU. Effects of low-intensity laser therapy on the orthodontic movement velocity of human teeth: a preliminary study. Lasers Surg Med. 2004;35(2):117-20. doi: 10.1002/lsm.20076. PMID 15334614
- [Background] Doshi-Mehta G, Bhad-Patil WA. Efficacy of low-intensity laser therapy in reducing treatment time and orthodontic pain: a clinical investigation. Am J Orthod Dentofacial Orthop. 2012 Mar;141(3):289-297. doi: 10.1016/j.ajodo.2011.09.009. PMID 22381489
- [Background] Heravi F, Moradi A, Ahrari F. The effect of low level laser therapy on the rate of tooth movement and pain perception during canine retraction. Oral Health Dent Manag. 2014 Jun;13(2):183-8. PMID 24984620
- [Background] Kau CH, Kantarci A, Shaughnessy T, Vachiramon A, Santiwong P, de la Fuente A, Skrenes D, Ma D, Brawn P. Photobiomodulation accelerates orthodontic alignment in the early phase of treatment. Prog Orthod. 2013 Sep 19;14:30. doi: 10.1186/2196-1042-14-30. PMID 24326198
- [Background] Nobrega C, da Silva EM, de Macedo CR. Low-level laser therapy for treatment of pain associated with orthodontic elastomeric separator placement: a placebo-controlled randomized double-blind clinical trial. Photomed Laser Surg. 2013 Jan;31(1):10-6. doi: 10.1089/pho.2012.3338. Epub 2012 Nov 15. PMID 23153291
- [Background] Tortamano A, Lenzi DC, Haddad AC, Bottino MC, Dominguez GC, Vigorito JW. Low-level laser therapy for pain caused by placement of the first orthodontic archwire: a randomized clinical trial. Am J Orthod Dentofacial Orthop. 2009 Nov;136(5):662-7. doi: 10.1016/j.ajodo.2008.06.028. PMID 19892282
- [Derived] AlSayed Hasan MMA, Sultan K, Ajaj M, Voborna I, Hamadah O. Low-level laser therapy effectiveness in reducing initial orthodontic archwire placement pain in premolars extraction cases: a single-blind, placebo-controlled, randomized clinical trial. BMC Oral Health. 2020 Jul 20;20(1):209. doi: 10.1186/s12903-020-01191-7. PMID 32690001